CLINICAL TRIAL: NCT06888583
Title: Fixation of Unstable Sacral Fractures by Transpedicular System
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Elsayed Elmoghany, Assistant Lecturer of Orthopaedic surgery, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Other Study IDs: 35358/3/22
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Fixation; Unstable Sacral Fractures; Transpedicular Sacral Fixation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transpedicular fixation group: Patients underwent transpedicular sacral fixation.
  Interventions: Procedure: Transpedicular fixation

INTERVENTIONS:
Procedure: Transpedicular fixation — Patients underwent transpedicular sacral fixation.

SUMMARY:
This research aimed to assess the role of the transpedicular Fixation system in the management of unstable sacral fractures in adults.

DETAILED DESCRIPTION:
Pelvic ring disruptions are high-energy injuries with a significant impact on quality of life and higher levels of mortality. Unstable sacral fracture is an unusual injury, and even though many studies implicate the surgical intervention as the treatment of choice, the purposes of surgery on sacral fractures include pelvic ring reconstruction, lumbopelvic stability restoration, fracture healing, early mobilization, fracture displacement prevention and improving the neurological deficiency. More and more surgeons are advocating for surgical management in the treatment of sacral fractures, and open reduction internal fixation (ORIF) has demonstrated marked benefits over conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years old age.
* Both sexes.
* Unstable AO sacral fracture type B and type C.
* Patient fit for surgery and hemodynamic stable patient.
* Closed fracture.

Exclusion Criteria:

* AO sacral fracture type A.
* Bedridden before the trauma.
* Patient unfit for surgery.
* Open sacral fractures.
* Sacral fractures with massive morel-lavallee lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective case series study was conducted on 21 patients with unstable sacral fractures at Tanta and Assiut University Hospitals from May 2022 to August 2024.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome | 1 year postoperatively
  Function results were assessed in terms of pain, standing and sitting, sexual function, and the need of assistance when walking, walking distance, and gait according to scoring system proposed by Majeed score. Five factors were assessed and scored: pain (30 points), standing (36 points), sitting (10 points), sexual intercourse (4 points) and work performance (20 points). The total score then gave a clinical grade as excellent (>85 points), good (70-84 points), fair (55-69 points) or poor (<55 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Elmoghany ME, Gharbo NO, Ayoub MA, Farouk OA, Mashal HEY. Fixation of unstable sacral fractures by transpedicular system: a prospective study. Int Orthop. 2025 Nov 14. doi: 10.1007/s00264-025-06673-3. Online ahead of print. PMID 41233652